CLINICAL TRIAL: NCT02804711
Title: A Phase Ia Single-center, Randomized, Double-blind, Placebo Controlled, Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of a Recombinant Staphylococcus Aureus Vaccine (Escherichia Coli) in Healthy Adults Aged 18-65 Years in China
Brief Title: A Clinical Trial to Evaluate a Recombinant Staphylococcus Aureus Vaccine (Escherichia Coli) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Chengdu Olymvax Biopharmaceuticals Inc. (Industry); Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT027
Record Dates: First submitted 2016-06-11; First posted 2016-06-17 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Staphylococcus Aureus Infection
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Four doses of low dose vaccine (Experimental): four doses of 15µg/0.6ml per dose
  Interventions: Biological: Low dosage of Staphylococcus aureus vaccine (15µg/0.6ml)
- Four doses of middle dose vaccine (Experimental): four doses of 30µg/0.6ml per dose
  Interventions: Biological: Middle dosage of Staphylococcus aureus vaccine (30µg/0.6ml)
- Four doses of high dose vaccine (Experimental): four doses of 60µg/0.6ml per dose
  Interventions: Biological: High dosage of Staphylococcus aureus vaccine (60µg/0.6ml)
- Three doses of low dose vaccine and one dose of placebo (Experimental): three doses of 15µg/0.6ml per dose and one dose of placebo
  Interventions: Biological: Low dosage of Staphylococcus aureus vaccine (15µg/0.6ml); Biological: Placebo
- Three doses of middle dose vaccine and one dose of placebo (Experimental): three doses of 30µg/0.6ml per dose and one dose of placebo
  Interventions: Biological: Middle dosage of Staphylococcus aureus vaccine (30µg/0.6ml); Biological: Placebo
- Three doses of high dose vaccine and one dose of placebo (Experimental): three doses of 60µg/0.6ml per dose and one dose of placebo
  Interventions: Biological: High dosage of Staphylococcus aureus vaccine (60µg/0.6ml); Biological: Placebo
- Four doses of placebo (Placebo Comparator): four doses of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dosage of Staphylococcus aureus vaccine (15µg/0.6ml)
  Arms: Four doses of low dose vaccine; Three doses of low dose vaccine and one dose of placebo
Biological: Middle dosage of Staphylococcus aureus vaccine (30µg/0.6ml)
  Arms: Four doses of middle dose vaccine; Three doses of middle dose vaccine and one dose of placebo
Biological: High dosage of Staphylococcus aureus vaccine (60µg/0.6ml)
  Arms: Four doses of high dose vaccine; Three doses of high dose vaccine and one dose of placebo
Biological: Placebo
  Arms: Four doses of placebo; Three doses of high dose vaccine and one dose of placebo; Three doses of low dose vaccine and one dose of placebo; Three doses of middle dose vaccine and one dose of placebo

SUMMARY:
Before this study, there will be an open-label, dose-escalation pilot study with a total of 30 participants with 10 per dosage group. The aim of the pilot study is to explore the preliminary safety of an experimental recombinant staphylococcus aureus vaccine.

This is a single center, double-blind, placebo control, dose-escalation phase 1 clinical trial. This study will determine the safety and side-effect profile, and immunogenicity of an experimental recombinant staphylococcus aureus vaccine. The study will be carried out following a dose-escalation method from the low dosage to the high dosage, i.e. the higher dosage vaccine could only be administrated after the first seven-day safety of the lower dosage vaccine is confirmed after safety observation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 65 years (aged over 18 and under 66 years).
* Able to comply with all clinical trial protocol requirements and willing to complete all the visit plan process during the whole clinical trial observation period.
* Able to understand the content of informed consent and willing to sign the informed consent.
* Able to complete the diary card independently.
* For females only (18-49 years), a negative urine pregnancy test and willing to practice continuous effective contraception during the study.
* Axillary temperature ≤37.0°C.

Exclusion Criteria:

First Immunization exclusion standard:

* Prior receipt of Staphylococcus aureus vaccine
* Any confirmed Staphylococcus aureus infection disease in the past 12 month.
* History of asthma, hereditary angioneurotic edema, diabetes, malignancy or other serious disease. Participation in the clinical trial is likely to increase the disease risk and interfere with the observation of clinical trial index.
* Prior blood donation or Blood loss over 400ml in the last 3 months;
* Coagulation disorders (coagulation factor deficiency, coagulopathy or platelet disorder) diagnosed by doctors, or obvious bruises or blood coagulation noticed.
* History of allergic disease likely to be exacerbated by any component of the vaccine, including allergy, urticaria, respiratory difficulty, angioneurotic edema or abdominal pain.
* Any autoimmune disease or immunodeficient state, parents, brother and sister with autoimmune disease or immunodeficient disease.
* Taking immunoglobulins and/or any blood products within the last 12 months.
* Asplenia, functional asplenia or asplenia caused by any situation or splenectomy.
* Any acute disease or acute attack of chronic disease in last 7 days.
* History of thyroidectomy or thyroid disease requiring treatment in the last 12 months.
* Immunosuppressor, cytotoxic therapy, inhaled corticosteroid (excluding corticosteroids spray treatment of allergic rhinitis, acute and non-concurrent corticosteroids treatment)
* Participation in another research study involving receipt of an investigational product in the last 30 days.
* Woman who is breast-feeding.
* Prior administration of attenuated vaccine in last 28 days.
* Prior administration of subunit vaccine, inactivated vaccine or allergic therapy in last 14 days.
* Current anti-tuberculosis prophylaxis or therapy
* Any other conditions may compromise the safety or availability of participants in the judgment of the investigator.

Following Immunization exclusion standard:

* Any grade 3 or more serious adverse reaction happen since the last vaccination.
* Other condition violates the inclusion criteria or meets the exclusion criteria is noticed after the first immunization.
* Acute or chronic infections at the vaccination day (axillary temperature>37.0°C).
* According to the investigator, the participant should not continue participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of injection site adverse reactions after vaccination | within 21 days after the vaccination
  Occurrence of solicited injection site adverse reactions within 21 days after vaccination with the Recombinant Staphylococcus aureus vaccine
Occurrence of systematic adverse reactions after vaccination | within 21 days after the vaccination
  Occurrence of solicited systematic adverse reactions within 21 days after vaccination with the Recombinant Staphylococcus aureus vaccine

SECONDARY OUTCOMES:
Occurrence of unsolicited adverse reactions after vaccination. | within 42 days after the vaccination
  Occurrence of unsolicited adverse reactions within 42 days after vaccination with the Recombinant Staphylococcus aureus vaccine
Occurrence of serious adverse events after the vaccination. | within 6 months after the vaccination
  Occurrence of serious adverse events within 6 months after the vaccination with the Recombinant Staphylococcus aureus vaccine
Changes of the blood routine after vaccination. | day 0-17 after the vaccination
  Changes of the blood routine after vaccination with the Recombinant Staphylococcus aureus vaccine on day 3, 7, 10, 14 and 17.
Changes of the blood biochemistry after vaccination. | day 0-17 after the vaccination
  Changes of the blood biochemistry after vaccination with the Recombinant Staphylococcus aureus vaccine on day 3, 7, 10, 14 and 17.
Geometric mean titre against specific antigens | within 6 months after the vaccination
  Geometric mean titre measured at day 0, 7, 14, 21, 42 and month 3, 6.
Geometric mean fold increase against specific antigens | within 6 months after the vaccination
  Geometric mean fold increase measured at day 7, 14, 21, 42 and month 3, 6.
Positive conversion rate of serum against specific antigens | within 6 months after the vaccination
  Positive conversion rate of serum measured at day 7, 14, 21, 42 and month 3, 6.

OTHER OUTCOMES:
Changes of the colonization of Staphylococcus aureus on nasal mucosus after vaccination. | within 6 months after the vaccination
  Changes of the colonization of Staphylococcus aureus on nasal mucosus after vaccination with the Staphylococcus aureus vaccine at day at day 3, 7, 10, 14, 17, 21, 42 and month 3, 6.
Specific functional antibody responses to the Staphylococcus aureus vaccine | within 6 months after the vaccination
  Specific functional antibody responses to the Staphylococcus aureus vaccine at day 7, 14, 21, 42 and month 3, 6.
Specific T cell immune responses to the Staphylococcus aureus vaccine. | within 6 months after the vaccination
  Specific T cell immune responses to the Staphylococcus aureus vaccine at day at day7, 14, 21, 42 and month 3, 6 measured by ELISpot.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaokui Hu, Taishing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu FC, Zeng H, Li JX, Wang B, Meng FY, Yang F, Gu J, Liang HY, Hu YM, Liu P, Peng LS, Hu XK, Zhuang Y, Fan M, Li HB, Tan ZM, Luo P, Zhang P, Chu K, Zhang JY, Zeng M, Zou QM. Evaluation of a recombinant five-antigen Staphylococcus aureus vaccine: The randomized, single-centre phase 1a/1b clinical trials. Vaccine. 2022 May 20;40(23):3216-3227. doi: 10.1016/j.vaccine.2022.04.034. Epub 2022 Apr 23. PMID 35473663